CLINICAL TRIAL: NCT01518491
Title: A Prospective, Randomized, Open Label Trial of NanoDOX™ Hydrogel Plus Vacuum Assisted Closure Therapy Versus Vacuum Assisted Closure Therapy Alone in Orthopedic Trauma Wounds.
Brief Title: Open Label Trial of NanoDOX Hydrogel in Orthopedic Trauma Wounds With and Without Vacuum Assisted Closure Therapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: NanoSHIFT LLC (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-DOX-NT/009
Record Dates: First submitted 2012-01-18; First posted 2012-01-26 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Orthopedic Trauma Wounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NanoDOX Hydrogel plus VAC (Experimental): NanoDOX™ Hydrogel in conjunction with serial wound debridement and irrigation on open traumatic orthopedic and soft tissue wounds in patients receiving negative pressure wound therapy/vacuum assisted closure (NPWT/VAC) with reticulated open cell foam (ROCF) dressings.
  Interventions: Drug: NanoDOX Hydrogel
- VAC Alone (Active Comparator): Serial wound debridement and irrigation alone in patients receiving negative pressure wound therapy/vacuum assisted closure (NPWT/VAC) with reticulated open cell foam (ROCF) dressings.
  Interventions: Other: VAC Alone

INTERVENTIONS:
Drug: NanoDOX Hydrogel — NanoDOX Hydrogel will be applied three time weekly to the wound for eight weeks along with VAC therapy
  Arms: NanoDOX Hydrogel plus VAC
Other: VAC Alone — Patients will receive VAC therapy three time weekly for eight weeks
  Arms: VAC Alone

SUMMARY:
The purpose of this study is to determine the effect of NanoDOX™ Hydrogel in conjunction with serial wound debridement and irrigation on the healing rates of open traumatic orthopedic and soft tissue wounds when compared to a serial wound debridement and irrigation alone in patients receiving negative pressure wound therapy/vacuum assisted closure (NPWT/VAC) with reticulated open cell foam (ROCF) dressings.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older
* Women of childbearing potential must have a negative urine pregnancy test at screening and at baseline
* Agree to use a double-barrier method of contraception during their participation in this study

  * condoms (with spermicide) and hormonal contraceptives OR
  * condoms (with spermicide) and intrauterine device OR
  * intrauterine device and hormonal contraceptives OR
* Abstains from sexual intercourse during their participation in this study
* Is with a same-sex partner and does not participate in bisexual activities where there is a risk of becoming pregnant
* Have a full-thickness trauma wound that is between 1.2cm2 and 24cm2 at initial screening
* Be able to apply study drug to their wound, or have a reliable and capable caregiver do it
* Subjects will have adequate blood flow to the wound as defined by transcutaneous oxygen tension (TcpO2) of >30mmHg recorded over intact epidermis at the wound margin.

Exclusion Criteria:

* Less than 18 years of age
* Pregnant or lactating woman or a female of childbearing potential who is not practicing acceptable form of birth control.
* Allergic to tetracycline, minocycline, demeclocycline, or any other known tetracycline derivative
* Tested positive for a doxycycline-resistant infection
* Have undergone treatment with systemic corticosteroid or immunosuppressive therapy in the past 2 months
* Currently undergoing dialysis for renal failure
* Have participated in another clinical research trial within the last 30 days
* Subject has wounds resulting from any cause other than trauma (diabetes, electrical burn, arterial insufficiency, chemical or radiation insult)
* Active or previous (within 60 days prior to the study screening visit) chemotherapy
* Active or previous (within 60 days prior to the study screening visit) radiation to the affected wound area to be treated by investigational drug or placebo
* Physical or mental disability or geographical concerns (residence not within reasonable travel distance) that would hamper compliance with required study visits
* The Investigator believes that the subject will be unwilling or unable to comply with study protocol requirements, including the shock wave treatment procedure, standard-of-care self-care requirements, and all study-related follow up visit requirements.
* History of sickle cell anemia
* History of infection with Human Immunodeficiency Virus
* History of other immunodeficiency disorders
* Severe anemia - Hgb < 7 g/dl (males) or < 6.5 (females)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2012-10 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Determine the effect of NanoDOX Hydrogel on the healing rates of open traumatic orthopedic wounds with and without vacuum assisted closure therapy. | participants will be followed for up to eight weeks
  To determine the effect of NanoDOX™ Hydrogel in conjunction with serial wound debridement and irrigation on the healing rates of open traumatic orthopedic and soft tissue wounds when compared to a serial wound debridement and irrigation alone in patients receiving negative pressure wound therapy/vacuum assisted closure (NPWT/VAC) with reticulated open cell foam (ROCF) dressings.

SECONDARY OUTCOMES:
Analyze the molecular changes in proinflammatory cytokine levels and bioburden that occur in traumatic orthopedic and soft tissue wounds | participants will have three visits per week for up to eight weeks
  Analyze the molecular changes in proinflammatory cytokine levels and bioburden (quantitative bacteriology and qRT-PCR for 16S rDNA) that occur in traumatic orthopedic and soft tissue wounds as a function of healing rate in the presence/absence of NanoDOX™ Hydrogel.

CONTACTS AND LOCATIONS:
Overall Officials: John Abernethy, MD, Study Director — Alachua Government Services, Inc.
Locations (2):
- United States (2):
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Univeristy of Missouri, Columbia, Missouri